CLINICAL TRIAL: NCT03015142
Title: Observational Clinical Study to Plan, Position and Check Instrument Placement for Spine Surgery Interventions
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY607-130099
Record Dates: First submitted 2017-01-02; First posted 2017-01-09 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Spinal Diseases
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- New image-guidance software: Patients in this group had spine surgery with new image-guidance software application.
  Interventions: Device: New image-guidance software

INTERVENTIONS:
Device: New image-guidance software — Patients in this group had spine surgery with new image-guidance software application

SUMMARY:
There is a clear need in spine surgery to place pedicle screws in the right place in the spine with good accuracy to avoid damage to important structures (spinal cord, nerve roots or vertebral arteries). The objective of the study was to investigate the accuracy of screw placement during spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject undergoing a spine surgery with pedicle screw placement
* Subject 16 years of age or older
* Subject able to give informed consent

Exclusion Criteria:

* Subject participating in a potentially confounding device or drug trial during the course of the study.
* Subject meeting an exclusion criteria according to national law (e.g. pregnant woman, breast feeding woman)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 16 years.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Elmi-Terander, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pedicle Screw Placement Using Augmented Reality Surgical Navigation with Intraoperative 3D Imaging. A First In-Human Prospective Cohort Study. — https://journals.lww.com/spinejournal/Abstract/publishahead/Pedicle_Screw_Placement_Using_Augmented_Reality.94855.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- New Image-guidance Software: Patients who had spine surgery with new image-guidance software.
Period: Overall Study
Arm/Group | New Image-guidance Software
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 9
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  Sweden | 21

OUTCOME MEASURES:

1. Primary Outcome: Clinical Accuracy of Pedicle Screw Placement Using New Image-guidance Software
Description: Clinical accuracy of pedicle screw placements using new image-guidance software assessed by three independent reviewers. Accuracy grading was done per Gertzbein classification.
  Gertzbein classification: grade 0 = breach 0 mm, grade 1 = breach < 2 mm, grade 2 = breach 2-4 mm, grade 3 = breach > 4 mm.
  Values in the data table represent the percentage of screw placements that were determined accurate by three independent reviewers.
Time Frame: During surgery, mean 6.71 hours
Population: 20 subjects were treated with the new image-guidance software. One was treated in the conventional method placing screws by free-hand method.
  Total of 253 screws (163 in thoracic, 77 in lumbar and 13 in sacral regions) were placed with new image-guidance software.
Measure: Number (95% Confidence Interval); unit: Percentage of screw placements
Units Other Than Participants: Screw placements
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Number analyzed (Screw placements) | 253
Percentage of screw placements | 94.1 [90.4 to 96.6]

2. Secondary Outcome: Procedure Time
Description: Time from skin incision to skin closure
Time Frame: During surgery, mean 6.71 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Hours | 6.71 (1.69)

3. Secondary Outcome: Time to Insert Pedicle Screw
Time Frame: Intraoperative, mean 5.18 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Minutes | 5.18 (4.03)

4. Secondary Outcome: Length of Hospitalization
Time Frame: From start of the interventional procedure until hospital discharge, approximately 5.3 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Days | 5.3 (1.71)

5. Secondary Outcome: System Usability Score (SUS Score)
Description: The SUS is a validated standard questionnaire to evaluate the system usability. Score varies between 0 and 100 (0 meaning the lowest usability score, 100 meaning highest usability score).
Time Frame: End of all surgeries
Population: Four independent physicians provided feedback via a validated system usability score (SUS)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 4
Scores on a scale | 75.6 (13.9)

6. Secondary Outcome: Patient Radiation Dose
Description: Radiation dose measured in Air Kerma (AK)
Time Frame: During surgery, mean 6.71 hours
Measure: Mean (Standard Deviation); unit: mGy (AK)
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
mGy (AK) | 158.60 (71.014)

7. Secondary Outcome: Patient Radiation Dose
Description: Radiation dose measured in Dose Area Product (DAP)
Time Frame: During surgery, mean 6.71 hours
Measure: Mean (Standard Deviation); unit: Gy.cm^2 (DAP)
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Gy.cm^2 (DAP) | 31.26 (12.604)

8. Secondary Outcome: Radiation Dose (Effective Dose) Received by Operator
Time Frame: During surgery, mean 6.71 hours
Population: There were 2 cases out of the 20 patients were the dosage information was missing.
Measure: Mean (Standard Deviation); unit: μSv
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 18
μSv | 0.21 (0.261)

9. Secondary Outcome: Procedure Related Complications
Description: Complication is leading to invasive intervention (e.g. blood sample, invasive intervention, IV/IM medication).
Time Frame: During surgery, mean 6.71 hours
Measure: Number; unit: Procedure related complications
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 20
Procedure related complications | 3

10. Secondary Outcome: Adverse Events, Adverse Device Effects and Device Deficiencies That Could Have Led to a Serious Adverse Event
Time Frame: From start of enrollment until hospital discharge, approximately 51 days
Population: 21 patients enrolled, 20 patients treated with new image-guidance software
Measure: Number; unit: Events
Groups:
- New Image-guidance Software: Patients who had spine surgery
Arm/Group | New Image-guidance Software
Number analyzed (Participants) | 21
Events
  Adverse Events (serious and non-serious) | 5
  Adverse Device Effects | 0
  Device deficiencies that could have led to SAE | 0

ADVERSE EVENTS:
Time Frame: From start of enrollment until hospital discharge, approximately 51 days
Arm/Group | New Image-guidance Software
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Image-guidance Software (N=20)
Pain right leg due to foramina stenosis by L5 screw. Screw was placed by free-hand. (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | New Image-guidance Software (N=20)
Horner's syndrome (Surgical and medical procedures) | 1 (1)
Postoperative pain (Surgical and medical procedures) | 1 (1)
Repeated Xper-CT (Surgical and medical procedures) | 1 (1)
Urticaria (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03015142/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT03015142/SAP_000.pdf